CLINICAL TRIAL: NCT03083366
Title: The Effectiveness of Early Sacral Nerve Stimulation in Improving Bladder- Related Complications and Quality of Life After Acute Traumatic Spinal Cord Injury
Brief Title: Sacral Nerve Stimulation in Improving Bladder Function After Acute Traumatic Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was unable to meet enrollment goals
Sponsor: University of Utah (Other)
Collaborators: Rancho Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Jeremy Myers, Associate Professor of Surgery, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 96153
Record Dates: First submitted 2017-01-27; First posted 2017-03-20 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injury, Acute; Neurogenic Bladder; Incontinence; Urinary Tract Infections
Keywords: spinal cord injury; Neurogenic; bladder; electrical stimulation; neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Randomized non-blinded study of sacral neuromodulation plus standard neurogenic bladder care versus standard neurogenic bladder care in patients with spinal cord injury
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sacral neuromodulation (Experimental): Bilateral sacral neuromodulation will start within 3 months of spinal cord injury, as well as standard neurogenic bladder care.
  Interventions: Device: PrimeAdvanced Surescan 97702 Neurostimulator - Medtronic (Minneapolis, MN)
- Standard care (No Intervention): Patients will receive standard neurogenic bladder care.

INTERVENTIONS:
Device: PrimeAdvanced Surescan 97702 Neurostimulator - Medtronic (Minneapolis, MN) — Bilateral s S3 sacral neuromodulation delivered via the PrimeAdvanced Surescan 97702 Neurostimulator - Medtronic (Minneapolis, MN)
  Other Names: Sacral neuromodulation
  Arms: Sacral neuromodulation

SUMMARY:
The purpose of this study is to see what effects sacral neuromodulation has on bladder function and quality of life in patients with acute spinal cord injury. Within 12-weeks of injury, participants will either receive an implanted nerve stimulator (like a pace-maker for the bladder) or standard care for neurogenic bladder. Patients will be assigned to one of these groups at random and followed for one year. The hypothesis is that early stimulation of the nerves will help prevent the development of neurogenic bladder.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Ability to implant device less than 12 weeks post-spinal cord injury (SCI)
* Presence of acute SCI at or above T12
* American Spinal Injury Association (ASIA) Scale A or B
* Expectation to perform clean intermittent catheterization (CIC) personally or have caretaker perform CIC

Exclusion Criteria:

* Inability to perform CIC
* Pre-existing SCI
* Pre-existing progressive neurological disorder
* Autonomic dysreflexia
* Prior sacral back surgery
* Posterior pelvic fracture with distortion of the sacroiliac joint
* Prior urethral sphincter or bladder dysfunction
* Chronic urinary tract infections prior to SCI
* Pregnancy at the time of enrollment
* Presence of coagulation disorder or need for anticoagulation that they cannot be stopped temporarily for procedure
* Any significant co-morbidity or illness that would preclude their participation or increase the risk to them having a surgical procedure
* Active untreated infection
* Traumatic injury to the genitourinary system
* Prior pelvic radiation, bladder cancer or other surgical procedure to the bladder that would effect baseline bladder physiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy B Myers, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Redshaw JD, Lenherr SM, Elliott SP, Stoffel JT, Rosenbluth JP, Presson AP, Myers JB; Neurogenic Bladder Research Group (NBRG.org). Protocol for a randomized clinical trial investigating early sacral nerve stimulation as an adjunct to standard neurogenic bladder management following acute spinal cord injury. BMC Urol. 2018 Aug 29;18(1):72. doi: 10.1186/s12894-018-0383-y. PMID 30157824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants from March 2019 to May 2022, with the first patient enrolled in August 2019. Patients were recruited from participating sites as well as online advertising.
Pre-assignment Details: There was a screening phase in order to identify eligible participants.
Period: Screening Period
Arm/Group | Sacral Neuromodulation | Standard Care
Started | 4 | 1
Completed | 3 | 1
Not Completed | 1 | 0
Not completed — Did not meet criteria (screen fail) | 1 | 0
Period: Enrollment Period
Arm/Group | Sacral Neuromodulation | Standard Care
Started | 3 | 1
Completed | 2 | 1
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacral Neuromodulation | Standard Care | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Cystometric Capacity
Description: Maximum bladder capacity as measured by urodynamic study at 12 months
Time Frame: 12 months
Population: All participants who completed the study. Data only collected for one participant in the sacral neuromodulation group at 12 months because the other did not return for their 12 month UDS. Data not collected for the participant in the standard of care group at 12 months because they did not return for their 12 month UDS.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 0
mL | 400 (0) |

2. Primary Outcome: Quality of Life Differences Measured by Mean SCI-QoL
Description: Participant-reported quality of life as assessed by the Spinal Cord Injury - Quality of Life (SCI-QOL) bladder question banks at 12 months. Scores range from 64-320 with a lower score indicating greater satisfaction with quality of life.
Time Frame: 12 months
Population: All participants who completed the study. Data only collected for one participant in the sacral neuromodulation group at 12 months because the other did not complete their 12 month questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
score on a scale | 130 (0) | 180 (0)

3. Primary Outcome: Number of Urinary Tract Infections Requiring Antibiotics
Time Frame: from enrollment through the end of follow-up at 12 months
Population: All enrolled participants.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 3 | 1
events | 5 | 2

4. Secondary Outcome: Maximum Cystometric Capacity at 3 Months
Description: Maximum bladder capacity as measured by urodynamic study at 3 months
Time Frame: 3 months
Population: All participants who completed the 3 month study visit. Data only collected for one participant in the sacral neuromodulation group at 3 months because the other did not return for their 3 month UDS.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
mL | 650 (0) | 231 (0)

5. Secondary Outcome: Bladder Compliance
Description: Bladder compliance as measured by urodynamic study (UDS) at 3 and 12 months.
Time Frame: 3, 12 months
Population: All participants who completed the 3 month study visit. Data only collected for one participant in the sacral neuromodulation group at 3 & 12 months because the other did not return for their 3 or 12 month UDS. Data not collected for the participant in the standard of care group at 12 months because they did not return for their 12 month UDS.
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
mL/cmH2O
  3 months | 25 (0) | 12.16 (0)
  12 months: number analyzed (Participants) | 1 | 0
  12 months | NA — Data collected was determined to be invalid due to grossly out of range value. |

6. Secondary Outcome: Presence of Detrusor Overactivity
Description: Presence of detrusor overactivity as evaluated by urodynamic study (UDS) at 3 and 12 months.
Time Frame: 3, 12 months
Population: as for outcome 5
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
events
  3 months | 0 | 1
  12 months: number analyzed (Participants) | 1 | 0
  12 months | 0 |

7. Secondary Outcome: Volume at First Detrusor Contraction
Description: Bladder volume at first detrusor contraction as measured by urodynamic study (UDS) at 3 and 12 months.
Time Frame: 3, 12 months
Population: All participants who completed the 3 month study visit. Data not collected for the sacral neuromodulation group at 3 & 12 months because one participant did not return for their 3 or 12 month UDS and this specific data point was inadvertently not recorded for the other participant during their 3 or 12 month UDS. Data not collected for the participant in the standard of care group at 12 months because they did not return for their 12 month UDS.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 0 | 1
mL
  3 months |  | 164 (0)
  12 months: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Pressure at First Detrusor Contraction
Description: Bladder pressure at first detrusor contraction as measured by urodynamic study (UDS) at 3 and 12 months.
Time Frame: 3, 12 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 0 | 1
cm H2O
  3 months |  | 16 (0)
  12 months: number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Daily Number of Catheterizations
Description: Daily number of catheterizations as reported in the participant diary.
Time Frame: 3, 6, 9, 12 months
Population: All participants who completed the 3 month study visit. Only one participant in the sacral neuromodulation group completed their diary entries, but did not complete the diary at 9 months. The participant in the standard care group did not complete this diary question at 6 or 12 months.
Measure: Mean (Standard Deviation); unit: catheterizations per day
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
catheterizations per day
  3 months | 4 (0) | 2 (0)
  6 months: number analyzed (Participants) | 1 | 0
  6 months | 3.67 (0) |
  9 months: number analyzed (Participants) | 0 | 1
  9 months |  | 6 (0)
  12 months: number analyzed (Participants) | 1 | 0
  12 months | 4 (0) |

10. Secondary Outcome: Average Catheterization Volume
Description: Average catheterization volume as determined by participant diary.
Time Frame: 3, 6, 9, 12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
mL
  3 months | 358.33 (0) | 461.67 (0)
  6 months: number analyzed (Participants) | 1 | 0
  6 months | 400 (0) |
  9 months: number analyzed (Participants) | 0 | 1
  9 months |  | 472.22 (0)
  12 months: number analyzed (Participants) | 1 | 0
  12 months | 79.42 (0) |

11. Secondary Outcome: Urinary Incontinence Episodes Per Day
Description: Urinary incontinence episodes per day as determined by participant diary.
Time Frame: 3, 6, 9, 12 months
Population: All participants who completed the 3 month study visit. Only one participant in the sacral neuromodulation group completed their diary entries, but did not complete the diary at 9 months. The participant in the standard care group did not complete this diary question at 3, 6, or 12 months.
Measure: Mean (Standard Deviation); unit: incontinence episodes per day
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
incontinence episodes per day
  3 months: number analyzed (Participants) | 1 | 0
  3 months | 0 (0) |
  6 months: number analyzed (Participants) | 1 | 0
  6 months | 0 (0) |
  9 months: number analyzed (Participants) | 0 | 1
  9 months |  | 0 (0)
  12 months: number analyzed (Participants) | 1 | 0
  12 months | 0 (0) |

12. Secondary Outcome: 24 Hour Pad Weight Test
Description: 24 hour pad weight as determined by participant diary.
Time Frame: 3, 6, 9, 12 months
Population: All participants who completed the 3 month study visit. Only one participant in the sacral neuromodulation group completed their diary entries, but did not complete the diary at 9 months. The participant in the standard care group did not complete this diary question at 6, 9, or 12 months.
Measure: Mean (Standard Deviation); unit: oz
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 1 | 1
oz
  3 months | 0 (0) | 0.81 (0)
  6 months: number analyzed (Participants) | 1 | 0
  6 months | 0 (0) |
  9 months: number analyzed (Participants) | 0 | 0
  12 months: number analyzed (Participants) | 1 | 0
  12 months | 0 (0) |

13. Secondary Outcome: Development of Hydronephrosis
Description: Development of hydronephrosis during the study period as determined by ultrasound at 12 months.
Time Frame: 12 months
Population: All participants who completed the study. Data not collected for either group because participants in both groups did not return for their 12 month ultrasound.
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Need for Anticholinergic Medication
Time Frame: from enrollment through the end of follow-up at 12 months
Population: All enrolled participants. Data not reported for one of the participants in the sacral neuromodulation group.
Measure: Count of Participants; unit: Participants
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

15. Secondary Outcome: Need for Onabotulinum Toxin A Injection
Time Frame: from enrollment through the end of follow-up at 12 months
Population: All enrolled participants. Data not reported for one of the participants in the sacral neuromodulation group.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 2 | 1
events | 1 | 1

16. Secondary Outcome: Need for Device Revision
Time Frame: from implant through the end of follow-up at 12 months
Population: All participants who had the device implanted were included.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 3 | 0
events | 0 |

17. Secondary Outcome: Device Explanation
Time Frame: from implant through the end of follow-up at 12 months
Population: All participants who had device implanted were included.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 3 | 0
events | 1 |

18. Secondary Outcome: Hospitalizations
Time Frame: from enrollment through the end of follow-up at 12 months
Population: All enrolled participants were included.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 3 | 1
events | 0 | 0

19. Secondary Outcome: Urologic Related Surgeries
Time Frame: from enrollment through the end of follow-up at 12 months
Population: All enrolled participants were included.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 3 | 1
events | 0 | 0

20. Secondary Outcome: Death
Time Frame: from enrollment through the end of follow-up at 12 months
Population: All enrolled participants were included.
Measure: Number; unit: events
Arm/Group | Sacral Neuromodulation | Standard Care
Number analyzed (Participants) | 3 | 1
events | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up period at 12 months
Description: Adverse events were collected via participant query, questionnaire, and laboratory testing.
Arm/Group | Sacral Neuromodulation | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacral Neuromodulation (N=3) | Standard Care (N=1)
Urinary tract infection (Renal and urinary disorders) | 2 (5) | 1 (2)

LIMITATIONS AND CAVEATS:
Target enrollment was not met and the study was terminated early. Due to the small number of subjects enrolled, there was insufficient data to achieve target power and statistically reliable results. Also, data were not collected for all participants at all study timepoints resulting in an incomplete dataset and uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03083366/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03083366/ICF_002.pdf